CLINICAL TRIAL: NCT06586957
Title: A Phase 1, First-in-human, Open-label Study to Evaluate the Safety, Tolerability, PK, and Preliminary Anti-tumor Activity of the Novel Oral CDK2 Degrader NKT3964 in Adults With Advanced/Metastatic Solid Tumors
Brief Title: A Study With NKT3964 for Adults With Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NiKang Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NKT3964-101
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor; Advanced Solid Tumor; Solid Tumor, Adult; Metastatic Tumor; Ovarian Cancer; Ovarian Neoplasms; Ovarian Carcinoma; Metastatic Ovarian Carcinoma; Endometrial Neoplasms; Endometrial Diseases; Metastatic Endometrial Cancer; Triple Negative Breast Cancer; Metastatic Endometrial Carcinoma; Advanced Endometrial Carcinoma; Advanced Ovarian Carcinoma; Gastric Cancer; Advanced Gastric Carcinoma; Metastatic Gastric Cancer; Metastatic Gastric Carcinoma; Small Cell Lung Cancer; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms; Platinum-resistant Ovarian Cancer; Platinum-refractory Ovarian Carcinoma; CCNE1 Amplification; Hormone Receptor Negative Breast Carcinoma; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Progesterone-receptor-positive Breast Cancer
Keywords: CDK 2 Inhibitor; CDK 4 Inhibitor; CDK 6 Inhibitor; CDK2 Degrader; Protein Degrader; PROTAC
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Diseases; Triple Negative Breast Neoplasms; Stomach Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Dose Escalation and Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation will assess the safety, efficacy, and PK/PD data of oral dosing NKT3964 at increasing dosage levels to determine the MTD and/or preliminary RDEs.
  Interventions: Drug: NKT3964
- Dose Expansion (Experimental): Dose expansion will include the RDE selected to determine the preliminary antitumor activity and the RP2D.
  Interventions: Drug: NKT3964

INTERVENTIONS:
Drug: NKT3964 — Oral CDK2 Degrader

SUMMARY:
The goal of the Dose Escalation phase of the study is to evaluate the safety, tolerability, pharmacokinetics (PK) and preliminary anti-tumor activity to determine the preliminary recommended dose for expansion (RDE) of NKT3964 in adults with advanced or metastatic solid tumors. The goal of the Expansion phase of the study is to evaluate the preliminary anti-tumor activity of NKT3964 at the RDE based on objective response rate (ORR) and determine the preliminary recommended Phase 2 dose (RP2D).

DETAILED DESCRIPTION:
Inclusion Criteria:

- Must have a pathologically confirmed, advanced and unresectable or metastatic solid tumor listed below with documented disease progression on last standard treatment.

For Part 1 only: Patients must be refractory to, or intolerant of existing therapy(ies) known to provide clinical benefit for their condition.

Part 1 Dose Escalation and Food Effect Sub-study:

1. Ovarian cancer
2. Endometrial cancer (only 'endometrioid' subtype requires CCNE1 amplification)
3. Gastric, gastroesophageal junction (GEJ) or esophageal adenocarcinoma with CCNE1 amplification
4. Small cell lung cancer (SCLC)
5. Triple-negative breast cancer (TNBC; HER2, estrogen receptor and progesterone receptor negative)
6. HR+ (includes estrogen-receptor or progesterone-receptor) and HER2- breast cancer (must have progressed following treatment with a CDK4/6 inhibitor, and is not suitable for endocrine therapy [ET])
7. Other solid tumors with CCNE1 amplification

Part 2 Dose Expansion:

Part 2A: HR+ and HER2- breast cancer that is locally advanced and unresectable (Stage III) or metastatic (Stage IV); previously treated with ≥1 line of SOC including CDK4/6 inhibitor plus ET and not suitable for further ET. Subjects must have progressed after receiving therapy for ≥3 months in the metastatic setting or for ≥6 months in the adjuvant setting. Subjects must have received ≤2 lines of systemic cytotoxic therapy (chemotherapy or cytotoxic antibody drug conjugate) in the metastatic setting.

Part 2B: Advanced platinum-based chemotherapy- resistant or refractory epithelial ovarian/fallopian/primary peritoneal carcinoma or clear cell ovarian cancer (defined as recurrence ≤6 months after completing platinum-based regimen) with progression on at least one platinum containing therapy and previously treated with ≤4 prior lines of systemic therapy administered for advanced/metastatic disease and with CCNE1 amplification.

Part 2C: Advanced unresectable or metastatic gastric, GEJ or esophageal adenocarcinoma with progression on at least one systemic therapy and previously treated with ≤3 prior lines of systemic therapy administered for advanced/metastatic disease, with CCNE1 amplification as determined by NGS by local liquid or tissue test.

Part 2D: Advanced endometrial adenocarcinoma or uterine papillary serous carcinoma previously treated with ≤4 prior lines of systemic therapy administered for advanced/metastatic disease with CCNE1 amplification.

Part 2E: Advanced/recurrent uterine carcinosarcoma previously treated with 1 prior platinum-based chemotherapy regimen and ≤3 prior lines of systemic therapy. Prior bevacizumab or PARP inhibitors are allowed and must be at least 3 weeks prior to the start of study drug.

* Measurable disease per RECIST v1.1, except for subjects with HR+/HER2- breast cancer or endometrial cancer (Part 1) who must have measurable or evaluable (including skin or bone lesion only) disease.
* Age ≥18 years
* ECOG PS 0-1
* Have adequate organ function
* Subjects with female reproductive organs must be surgically sterile, post-menopausal, or, if of child-bearing potential, must meet pre-specified criteria
* Subjects who are capable of insemination must meet pre-specified criteria
* Ability to swallow oral medications.
* Consent to provide archived tumor tissues and paired tumor biopsy at pretreatment and on-treatment.

Exclusion Criteria:

* Locally advanced solid tumor that is a candidate for curative treatment through radical surgery and/or radiotherapy, or chemotherapy.
* History of another malignancy with exceptions
* History of lymphohistiocytic or lymphoid hyperplasia; hemophagocytic lymphohistiocytosis.
* Failed to recover from effects of prior anticancer treatment therapy to baseline or Grade ≤ 1 severity (per CTCAE)
* Clinically significant cardiovascular event within 6 months prior to start of NKT3964 treatment
* Known active CNS metastases and/or carcinomatous meningitis
* Clinically active interstitial lung disease currently requiring treatment
* History of uveitis, retinopathy or other clinically significant retinal disease
* Active or chronic corneal disorders, other active ocular conditions requiring ongoing therapy, or any clinically significant corneal disease
* Active wound healing from major surgery within 1 month or minor surgery within 10 days before the first dose of NKT3964.
* Known human immunodeficiency virus (HIV), active hepatitis B or C infection
* Prior investigative treatment with a selective or nonselective CDK2 inhibitor or degrader
* Childs-Pugh class B or C cirrhosis or any other clinically significant liver disorder
* Palliative radiation therapy within 14 days or other radiation therapy within 4 weeks prior to C1D1

ELIGIBILITY:
Inclusion Criteria:

- Must have a pathologically confirmed advanced and unresectable or metastatic solid tumor listed below with documented disease progression on last standard treatment. Part 1 only: subjects must be refractory to, or intolerant of existing therapy(ies) known to provide clinical benefit for their condition.

Dose Escalation:

1. Ovarian cancer
2. Endometrial cancer (only endometrioid subtype will require CCNE1 amplification)
3. Gastric, gastroesophageal junction (GEJ) or esophageal adenocarcinoma with CCNE1 amplification
4. Small cell lung cancer (SCLC)
5. Triple-negative breast cancer (TNBC; HER2, estrogen receptor and progesterone receptor negative)
6. HR+ (includes estrogen-receptor or progesterone-receptor) and HER2- breast cancer (must have progressed following treatment with a CDK4/6 inhibitor, and is not suitable for endocrine therapy [ET])
7. Other solid tumors with CCNE1 amplification

Dose Expansion:

Part 2A: HR+ and HER2- breast cancer that is locally advanced and unresectable (Stage III) or metastatic (Stage IV); previously treated with ≥1 line of standard of care (SOC) including CDK4/6 inhibitor plus ET and not suitable for further ET. Subjects must have progressed after receiving therapy for ≥3 months in the metastatic setting or for ≥6 months in the adjuvant setting. Subjects must have received ≤2 lines of systemic cytotoxic therapy (chemotherapy or cytotoxic antibody drug conjugate [ADC]) in the metastatic setting..

Part 2B: Advanced platinum-based-chemotherapy resistant or refractory epithelial ovarian/fallopian/primary peritoneal carcinoma or clear cell ovarian cancer (defined as recurrence ≤6 months after completing platinum-based regimen) with progression on at least one platinum containing therapy and previously treated with ≤4 prior lines of systemic therapy administered for advanced/metastatic disease and with CCNE1 amplification.

Part 2C: Advanced unresectable or metastatic gastric, GEJ or esophageal adenocarcinoma with progression on at least one systemic therapy and previously treated with ≤3 prior lines of systemic therapy administered for advanced/metastatic disease, with CCNE1 amplification as determined by NGS by local liquid or tissue test.

Part 2D: Advanced endometrial adenocarcinoma or uterine papillary serous carcinoma previously treated with ≤4 prior lines of systemic therapy administered for advanced/metastatic disease with CCNE1 amplification.

Part 2E: Advanced/recurrent uterine carcinosarcoma previously treated with 1 prior platinum-based chemotherapy regimen and ≤3 prior lines of systemic therapy. Prior bevacizumab or PARP inhibitors are allowed and must be at least 3 weeks prior to the start of study drug.

* Have adequate organ function
* Subjects with female reproductive organs must be surgically sterile, post-menopausal, or must be willing to use highly effective method(s) of contraception
* Ability to swallow oral medications.
* Consent to provide archived tumor tissues and paired tumor biopsy at pretreatment

Exclusion Criteria:

* Locally advanced solid tumor that is a candidate for curative treatment through radical surgery and/or radiotherapy, or chemotherapy.
* History of another malignancy with exceptions
* History of lymphohistiocytic or lymphoid hyperplasia; hemophagocytic lymphohistiocytosis.
* Failed to recover from effects of prior anticancer treatment therapy to baseline or Grade ≤ 1 severity (per CTCAE)
* Clinically significant cardiovascular event within 6 months prior to start of NKT3964 treatment
* Known active CNS metastases and/or carcinomatous meningitis
* Active interstitial lung disease currently requiring treatment
* History of uveitis, retinopathy or other clinically significant retinal disease
* Active or chronic corneal disorders, other active ocular conditions requiring ongoing therapy, or any clinically significant corneal disease
* Active wound healing from major surgery within 1 month or minor surgery within 10 days before the first dose of NKT3964.
* Known human immunodeficiency virus (HIV), active hepatitis B or C infection
* Prior investigative treatment with a selective or nonselective CDK2 inhibitor or degrader
* Childs-Pugh class B or C cirrhosis or any other clinically significant liver disorder
* Palliative radiation therapy within 14 days or other radiation therapy within 4 weeks prior to C1D1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) events | 28 Days
  DLTs graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Objective Response Rate (ORR) | 1 Year
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as determined by the Investigator

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 Year
  PFS defined as the time from the date the participant started study drug to the date the participant experiences an event of disease progression or death.
Duration of Response (DOR) | 2 Year
  Duration of overall response is defined as the time from the date of first confirmed CR or PR, assessed by investigator and based on RECIST v. 1.1, to the documented date of progressive disease (PD) including clinical progression, or death due to any cause, or the start of subsequent anticancer therapy, whichever occurred first.
Disease control rate | 1 Year
  Disease control rate defined as CR + PR + stable disease [SD] for at least 8 weeks
Overall Survival (OS) | 2 Year
  OS defined as the time from the date the participant started study drug to death for any reason.
Time to Response (TTR) | 1 Year
  TTR is defined as the time from first dose to the first documented CR or PR which is subsequently confirmed.
Number of Participants with Adverse Events | 2 Year
  An adverse event (AE) is defined as any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related.
Maximum observed plasma concentration (Cmax) of NKT3964 with and without a high-fat and/or low-fat meal | 1 Month
  Maximum observed plasma concentration (Cmax) of NKT3964
Time to maximum observed plasma concentration of NKT3964 (Tmax) with and without a high-fat and/or low-fat meal | 1 Month
  Time to maximum observed plasma concentration of NKT3964 (Tmax)
Observed trough concentration of NKT3964 (Ctrough) | 88 Weeks
  Observed trough concentration of NKT3964 (Ctrough)
Area under the plasma concentration-time curve (AUC0-t) of NKT3964 with and without a high-fat and/or low-fat meal | 1 Month
  Area under the plasma concentration-time curve (AUC0-t) of NKT3964
Apparent clearance (CL/F) of NKT3964 | 1 Month
  Apparent clearance (CL/F)
Apparent volume of distribution (V/F) of NKT3964 | 1 Month
  Apparent volume of distribution (V/F)
Half-life (t1/2) of NKT3964 | 1 Month
  Half-life (t1/2)
Accumulation ratio (AR) of NKT3964 | 1 Month
  Accumulation ratio (AR)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Arkansas Medical School, Little Rock, Arkansas
  - University of California - Los Angeles, Los Angeles, California
  - UCSF, San Francisco, California
  - SCRI at HealthOne, Denver, Colorado
  - Florida Cancer Specialists & Research Institute, Lake Mary, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Kansas, Fairway, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Sidney Kimmell Cancer Center - Jefferson Health, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee
  - NEXT Oncology, Austin, Texas
  - UT Southwestern, Dallas, Texas
  - Intermountain Health, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
IPD are not planned to be shared at this time